CLINICAL TRIAL: NCT02296164
Title: A PROspective, Observational, US-based Study Assessing Outcomes, Adverse Events, Treatment Patterns, and Quality of Life in Patients Diagnosed With Mycosis Fungoides Cutaneous T-cell Lymphoma and Treated With Valchlor®
Brief Title: Clinical Study Assessing Outcomes, Adverse Events, Treatment Patterns, and Quality of Life in Patients Diagnosed With Mycosis Fungoides Cutaneous T-cell Lymphoma
Acronym: PROVe
Status: Completed | Type: Observational
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-079A501
Record Dates: First submitted 2014-11-07; First posted 2014-11-20 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Mycosis Fungoides
Keywords: PROVe; CTCL; Mechlorethamine; Cutaneous T-cell lymphoma; Mycosis fungoides cutaneous T-cell lymphoma; Valchlor; Dermatology; MF-CTCL; Mycosis Fungoides; Oncology
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Neoplasms | interventions — Amines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MF-CTCL Patients receiving Valchlor: Patients will undergo clinical assessments and receive standard medical care, as determined by the patients' physician, in the real world setting. With the exception of protocol-required patient completed questionnaires for symptoms and Quality Of Life.
  Interventions: Drug: Valchlor

INTERVENTIONS:
Drug: Valchlor — Valchlor gel 0.016%
  Other Names: Mechlorethamine gel

SUMMARY:
The Valchlor PROVe study is a multi-center, prospective, observational, US-based drug study that longitudinally follows patients with Mycosis Fungoides Cutaneous T-cell Lymphoma (MF-CTCL) who are receiving therapy with Valchlor. Patients will be followed prospectively for a maximum of 2 years from the date of signed informed consent (enrollment) until end of study. Continuation in the study is not contingent on continuation of Valchlor.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational, US-based drug study. All consecutive Mycosis Fungoides Cutaneous T-cell Lymphoma (MF-CTCL) patients being treated with Valchlor will be invited to enroll in this study.Patients will undergo clinical assessments and receive standard medical care, as determined by the patients' physician, in the real world setting. With the exception of protocol-required patient completed questionnaires for symptoms and QOL, there are no specific or mandated clinical assessments to be performed. Patients will be followed prospectively for a maximum of 2 years

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years of age) diagnosed with MF CTCL and being treated with Valchlor. This includes patients newly initiating Valchlor OR patients continuing treatment with Valchlor:

  * Patients newly initiating Valchlor are patients who have their first office visit after having initiated Valchlor.
  * Patients continuing treatment with Valchlor includes patients who are actively taking Valchlor on the day of enrollment.
* Signed patient informed consent.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Bailey, Study Director — Helsinn Therapeutics (U.S.), Inc
Locations (31):
- United States (31):
  - Investigator Site, Little Rock, Arkansas
  - Investigator Site, Duarte, California
  - Investigator Site, La Mesa, California
  - Investigator Site, San Francisco, California
  - Investigator Site, Santa Ana, California
  - Investigator Site, Aurora, Colorado
  - Investigator Site, New Haven, Connecticut
  - Investigator Site, Coral Gables, Florida
  - Investigator Site, Hollywood, Florida
  - Investigator Site, Naples, Florida
  - Investigator Site, Tampa, Florida
  - Investigator Site, Atlanta, Georgia
  - Investigator Site, Chicago, Illinois
  - Investigator Site, New Orleans, Louisiana
  - Investigator Site, Boston, Massachusetts
  - Investigator Site, Ann Arbor, Michigan
  - Investigator Site, Jackson, Mississippi
  - Investigator Site, St Louis, Missouri
  - Investigator Site, Henderson, Nevada
  - Investigator Site, East Windsor, New Jersey
  - Investigator Site, Brooklyn, New York
  - Investigator Site, Fairport, New York
  - Investigator Site, New York, New York
  - Investigator Site, The Bronx, New York
  - Investigator Site, Cleveland, Ohio
  - Investigator Site, Exton, Pennsylvania
  - Investigator Site, Philadelphia, Pennsylvania
  - Investigator Site, Pittsburgh, Pennsylvania
  - Investigator Site, Charleston, South Carolina
  - Investigator Site, Dallas, Texas
  - Investigator Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
observational study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study registered 301 consecutive adult patients (Only registered/not enrolled:1; Enrolled: 300) diagnosed with MF-CTCL and being treated with Valchlor, regardless of other MF-CTCL therapies received before or at enrollment. All patients were enrolled from 46 participating centers/clinics in university-affiliated or community hospitals in the US
Pre-assignment Details: All consecutive MF-CTCL patients being treated with Valchlor were invited to enroll in this study. Two patients were not eligible as they were not on Valchlor at time of study start
Groups:
- MF-CTCL Patients Receiving Valchlor: Patients will undergo clinical assessments and receive standard medical care, as determined by the patients' physician, in the real world setting. With the exception of protocol-required patient-completed questionnaires for symptoms and QOL, there were no specific or mandated clinical assessments performed, and patients did not receive experimental intervention or treatment as a consequence of their participation in this study. Continuation in the study was not contingent on continuation of Valchlor.
  Valchlor: Valchlor gel 0.016%
Period: Overall Study
Arm/Group | MF-CTCL Patients Receiving Valchlor
Started (Registered: 301; Only registered/not enrolled:1; Enrolled: 300) | 298 (2 patients not eligible as were not on Valchlor at time of study start)
Completed | 188
Not Completed | 110

BASELINE CHARACTERISTICS:
Arm/Group | MF-CTCL Patients Receiving Valchlor
Number analyzed (Participants) | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 162
  >=65 years | 136
Sex: Female, Male [Count of Participants; unit: Participants] — Adult Males and Females
  Participants
    Female | 119
    Male | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11
  African American | 45
  Hispanic or Latino | 29
  Asian | 2
  Native Hawaiian/other Pacific Islander | 6
  Unknown or ≥2 races/ethnicities | 2
  Not Disclosed | 203
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 298
diagnosed with MF-CTCL and being treated with Valchlor. [Count of Participants; unit: Participants] | 298

OUTCOME MEASURES:

1. Primary Outcome: Treatment Responders Using Body Surface Area (BSA) at 12 Months
Description: The primary efficacy endpoint was the proportion of patients who are responders to treatment at the 12-month timepoint using a ≥50% reduction from baseline in BSA as the definition of a responder in the group of patients who used mechlorethamine plus corticosteroids and possibly another treatment.
Time Frame: 12 Months
Population: The primary efficacy endpoint was the proportion of patients who are responders to treatment at the 12-month timepoint using a ≥50% reduction from baseline in BSA as the definition of a responder in the group of patients who used mechlorethamine plus corticosteroids and possibly another treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MF-CTCL Patients Receiving Valchlor
Number analyzed (Participants) | 298
Participants | 44

ADVERSE EVENTS:
Time Frame: The definition of an on-study event is one that occurs on the day of enrollment or later, but before the date of study discontinuation or completion ( 2 years).
Description: The frequency and percentage of patients experiencing any on-study Adverse Events (AEs), Serious Adverse Events (SAEs), or death.
  Additional detail for Adverse Events (AEs) of special interest (e.g., dermatitis).
  Serious Adverse Events (SAEs) both including and excluding events that were not concurrent with Valchlor exposure.
Arm/Group | MF-CTCL Patients Receiving Valchlor
All-Cause Mortality (participants affected / at risk) | 0/298
Serious Adverse Events (participants affected / at risk) | 23/298
Other Adverse Events (participants affected / at risk) | 104/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF-CTCL Patients Receiving Valchlor (N=298)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer with HLT skin neoplasm malignant and unspecified (exc. Melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Packed red blood cell transfusion (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF-CTCL Patients Receiving Valchlor (N=298)
Dermatitis (Skin and subcutaneous tissue disorders) | 38 (38)
Erythema (Skin and subcutaneous tissue disorders) | 15 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (29)
Skin irritation (Skin and subcutaneous tissue disorders) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT02296164/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02296164/SAP_002.pdf